CLINICAL TRIAL: NCT06850584
Title: A Confirmatory Study of the Simplified Chinese Version of the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) Battery (2nd Edition) to Assess Cognitive Impairment in Patients with Traumatic Brain Injury
Brief Title: Validation Study of Simplified Chinese Version of LOTCA Scale in the Assessment of Cognitive Impairment in Patients with Traumatic Brain Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing Broad Biopharmaceutical Ltd. (Network)
Responsible Party: Sponsor
Other Study IDs: LOTCA-YZ-1
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group
  Interventions: Other: Observation
- Control group
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — The study was observational and did not involve any intervention.

SUMMARY:
In this study, 300 patients aged ≥18 years old with traumatic brain injury (case group) and hospitalized patients without central nervous system disease or their family members and accompanying staff (control group) were selected as the study objects. At baseline, participants completed the Mini-mental State Examination (MMSE), the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery, the Glasgow Coma Scale (GCS), and the Alzheimer's Disease Rating Scale Cognitive Subscale (ADAS-Cog11). The evaluation process of the first LOTCA test was videotaped by a person. 2 weeks after the evaluation, the same two scale raters watched the video and rated it independently again. After 3 months, the subjects completed MMSE, LOTCA battery, GCS, ADAS-Cog11 assessment again.

ELIGIBILITY:
Inclusion Criteria:

- Case group: Patients with traumatic brain injury

Inclusion Criteria:

1. Age> = 18 years old, male or female;
2. patients with traumatic brain injury;
3. The Mini-Mental State Examination (MMSE) score was lower than normal, and the cut-off value for diagnosis was determined according to different education levels: illiteracy (uneducated) <=19 points, primary school level <=22 points, junior high school level and above < = 26 points;
4. Voluntary participation and ability to complete the study and sign the informed consent form in accordance with the requirements of the study protocol.

Control group: family members or accompanying persons of patients in the same period

Inclusion Criteria:

1. Age> = 18 years old, male or female;
2. recent emotional stability;
3. Mini-Mental State Examination (MMSE) score was normal;
4. Voluntary participation and ability to complete the study and sign the informed consent form in accordance with the requirements of the study protocol.

Exclusion Criteria:

- Case group: Patients with traumatic brain injury

Exclusion Criteria:

1. The study subject is in a lethargic state, coma, or persistent vegetative state;
2. the disease progresses rapidly or is accompanied by serious complications;
3. The subject has severe language dysfunction or/or bilateral upper limb motor function loss;
4. the study subject has severe visual and/or hearing impairment;
5. The subject has a severe mental disorder, physical weakness or other conditions (such as intolerance to the test or uncooperation, etc.);
6. Those who have a history of drug abuse within 6 months before screening or those who have used drugs within 3 months before screening;
7. Those who are considered by the investigator to be unsuitable to participate in this study or cannot complete this study for other reasons.

Control group: family members or accompanying persons of patients in the same period

Exclusion Criteria:

1. History of congenital or acquired central nervous system disease (including history of traumatic brain injury, cerebrovascular accident, etc.);
2. Those who have a history of drug abuse within 6 months before screening or who have used drugs within 3 months before screening;
3. Those who are considered by the investigator to be unsuitable to participate in this study or cannot complete this study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age ≥18 years old, male or female, patients with traumatic brain injury (case group) and family members or caregivers of patients at the same time (control group).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluator Reliability of the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery | At baseline
Retest Reliability of the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery | 2 weeks Later
Internal Consistency Reliability of the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery | At baseline
Content Validity of the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery | At baseline
Construct Validity of the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery | At baseline
Discriminative Validity of the Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery | At baseline
The change of Loewenston Occupational Therapy Cognitive Assessment (LOTCA) battery score from baseline values | 3 months later
The change of Alzheimer's Disease Assessment Scale - Cognitive Subscale 11 score from baseline values | 3 months later
Correlation between LOTCA score change from baseline and ADAS-Cog11 score change from baseline | 3 months later
The area under ROC curve and the sensitivity, specificity and Jorden index under optimal threshold of LOTCA score change from baseline value | 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: tong ru Yu, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (4):
- China (4):
  - The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huaian, Jiangsu
  - Suzhou Jiulong Hospital, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No